CLINICAL TRIAL: NCT02573246
Title: Neuromodulation Enhanced Cognitive Restructuring: A Proof of Concept Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00066383
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Results first posted 2021-05-10 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-05

CONDITIONS: Anxiety; Depression; Personality Disorders; Trauma and Stress-related Disorders; Somatic Disorders; Obsessive Compulsive Disorders; Eating Disorders; Difficulties With Cognitive Emotion Regulation
Keywords: neurostimulation; cognitive restructuring; TMS; emotion regulation; MRI; Emotional Memory Task; Reappraisal; Distraction
MeSH Terms: conditions — Anxiety Disorders; Depression; Personality Disorders; Trauma and Stressor Related Disorders; Compulsive Personality Disorder; Feeding and Eating Disorders; Emotional Regulation | interventions — Cognitive Restructuring

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of 2 studies (main and supplement) that ran concurrently. 83 participants were enrolled in the main study, and 65 in the supplement.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Restructuring+rTMS (left) (Experimental): Participants in this arm will be administered the neuromodulation enhanced cognitive restructuring intervention over the left side of the brain and will partake in short term and long term follow up testing.
  Interventions: Behavioral: Cognitive Restructuring; Device: rTMS
- Cognitive Restructuring + sham rTMS (Sham Comparator): Participants in this arm will receive cognitive restructuring alone as an active intervention and will partake in short term and long term follow up testing.
  Interventions: Behavioral: Cognitive Restructuring; Device: Sham rTMS
- Cognitive Restructuring+rTMS (right) (Experimental): Participants in this arm will be administered the neuromodulation enhanced cognitive restructuring intervention over the right side of the brain and will partake in short term and long term follow up testing.
  Interventions: Behavioral: Cognitive Restructuring; Device: rTMS

INTERVENTIONS:
Behavioral: Cognitive Restructuring — Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.
Device: rTMS — rTMS is a neurostimulation intervention where the participant receives 15 minutes of high frequency (10 HZ) transcranial magnetic stimulation pulses
  Arms: Cognitive Restructuring+rTMS (left); Cognitive Restructuring+rTMS (right)
Device: Sham rTMS — Sham rTMS is a placebo intervention aimed to mimic the effects of repetitive transcranial magnetic stimulation with no known direct benefit for the participant.
  Arms: Cognitive Restructuring + sham rTMS

SUMMARY:
Psychological treatments are effective, but take a long time and can be burdensome. Therefore, avenues to optimize behavioral treatments are needed. Despite important advancements, neuroscience has had a limited effect on psychotherapy development. Therefore, one paradigm shift would be to develop neuroscience informed behavioral treatments.

The investigators identified from the literature a problem that affects several mental disorders (emotion dysregulation) and a neural circuit that underlies this important concern. They found that this circuit is dysfunctional in those with psychopathology but can be changed with treatment. The goal is in one session to train this brain network to operate more efficiently and to test the short and long term effects of this intervention. The investigators plan to engage this brain network using a traditional psychotherapy strategy (cognitive restructuring) and to enhance learning using repetitive transcranial magnetic stimulation (rTMS), a neuromodulation technique through which magnetic stimulation enhances the electrical activity in brain areas close to the scalp.

The study team proposed two studies to examine this novel approach, In one of the studies 83 participants were enrolled and 47 eligible participants were divided into 3 groups. All participants were trained in emotion regulation by first being asked to remember an event where they experienced a negative emotion and then being instructed either to think differently about the event, or to wait. Participants simultaneously underwent either active (left or right side of brain) or sham rTMS. In a second study 65 participants were enrolled, and 31 were assigned to either active left or sham rTMS guided using neuroimaging results. Across both studies, the investigators measured regulation in the lab and during a-week long naturalistic assessment. Participants in the second study returned for a follow up neuroimaging visit at the end of this week. Participants returned for a one moth follow up assessment and to rate feasibility, acceptability, and provide feedback. This proof of concept set of studies demonstrated feasibility and preliminary efficacy for this approach, which opens new frontiers for neuroscience informed treatment development.

DETAILED DESCRIPTION:
Despite significant advancements in psychiatric research, the majority of adults with mental health disorders do not benefit from current evidence-based treatments, especially if they have difficulties managing negative emotions. One solution to this unmet clinical need is to take a neuroscience-informed approach to treatment development in order to radically change patient care. Despite an explosion of research on the neurobiological underpinnings of emotion, emotion regulation, and psychopathology, there have been few attempts to use such findings to advance behavioral treatments. Neuroscience-informed treatment development could optimize psychotherapy gains and reduce burden on therapists and clients. Therefore, we propose to build a fundamentally novel approach to treating difficulties managing negative emotions (or emotion dysregulation) that builds on the strength of current therapies, but that also accelerates and enhances gains.

Adults with several different psychiatric disorders have difficulty managing negative emotions, a problem that has been traced back to impairments in the fronto-limbic brain circuitry. In healthy samples this neural network is activated in response to tasks requiring regulation of emotional arousal and disrupting this circuit leads to psychiatric symptoms. In psychiatric samples, this circuit is underperforming as evidenced by (1) hyperactivity in the amygdala (the brain structure that signals emotional arousal), (2) slow return to baseline after amygdala activation, (3) hypoactivity in frontal regions (responsible for regulation), and (3) insufficient cross-talk between these regions when patients experience negative emotional arousal. Evidence-based cognitive-behavioral psychotherapy and neurostimulation are two different interventions that can remediate function in impaired brain circuits. Both interventions have evidence of success in changing the fronto-limbic network but also need improvement. Therefore, the investigators plan to combine magnetic brain stimulation and cognitive restructuring (an evidence-based behavioral treatment for difficulties managing emotions) in a one-session intervention.

The investigators recruited participants for two studies. In one study, 83 transdiagnostic adults (i.e., who meet criteria for any DSM 5 disorder) who engage in cognitive restructuring with low frequency as measured by an established questionnaire were enrolled and 47 were randomly assigned to either active (left or right) or sham repetitive transcranial magnetic stimulation (rTMS). In a second study, 65 transdiagnostic adult participants with high emotional dysregulation were enrolled, and 31 were randomly assigned to active left or sham rTMS guided using neuroimaging analyses. All included participants practiced reducing negative emotions (induced with standardized autobiographical stressors) using cognitive restructuring while undergoing high frequency or sham rTMS to the right or left dorsolateral prefrontal cortex. Standardized, established procedures were used to teach cognitive restructuring, to generate personalized stressors, to induce negative emotional arousal, and to implement the one session of rTMS. Immediate effects were evaluated using measures of emotional arousal and regulation during the intervention and for one week afterwards using 8 daily automated mobile phone calls. Long-term effects in emotion regulation, functional and psychiatric impairment were examined at 1-week and 1-month follow-up interviews.

Participants in the imaging portion of the study underwent an MRI before the intervention day. This imaging session included training in the emotion regulation task to be performed in the scanner, including practice in reappraisal and distraction; a memory cue assessment to rehearse cuing of memories; a mock scan if necessary, MRI safety screening confirmation, structural (Diffusion tensor imaging and anatomical) and functional MRI (fMRI) images will be collected. During the fMRI scan, participants completed the emotional regulation task where they were asked to recall an emotional memory from the Emotional Memory selection tasks and then be cued to reappraise, distract or allow negative emotions. At the end of the trials, participants rated their current emotional state. At the one week follow up, in addition to the tasks described above, they returned to complete a second MRI after 1 week where they were reoriented to the emotion regulation task, had structural and functional MRI images collected with the emotion regulation task occurring during the fMRI portion.

The investigators hypothesized that rTMS would enhance cognitive restructuring by yielding a quicker reduction in emotional arousal when compared to sham TMS, and would lead to more frequent use of the cognitive restructuring in the natural environment. This set of studies is intended to launch a series of investigations using innovative paradigms to optimize treatments for psychiatric disorders and it could lead to the next generation of neuroscience-informed behavioral interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Has difficulty thinking differently in emotional situations
2. Meets diagnostic criteria for a current DSM-5 depressive, anxiety, obsessive-compulsive, somatic, personality, eating, or trauma and stress-related disorders (including in partial remission): major depressive disorder, persistent depressive disorder, panic disorder, agoraphobia, social anxiety disorder, specific phobia, generalized anxiety disorder, obsessive-compulsive disorder, trichotillomania, excoriation disorder, hoarding disorder, body dysmorphic disorder, other specified, or unspecified obsessive-compulsive disorder, posttraumatic stress disorder, acute stress disorder, adjustment disorders, somatic symptom disorder, conversion disorder, anorexia nervosa, bulimia nervosa, binge-eating disorder, borderline personality disorder, narcissistic personality disorder, histrionic personality disorder, antisocial personality disorder, paranoid personality disorder, schizoid personality disorder, schizotypal personality disorder, avoidant personality disorder, dependent personality disorder, obsessive-compulsive personality disorder, personality disorder unspecified, depressive disorder unspecified, anxiety disorder unspecified.
3. Willing and able to participate in the intervention and all required study visits, stay on the same dose of psychiatric medication (if any) throughout the study, not participate in cognitive-behavioral therapy throughout their participation in the study.
4. Has cellphone that can be used during the ambulatory assessment portion of the study.

Exclusion Criteria:

1. Current or recent (within the past 6 months) substance dependence disorder(excluding nicotine and caffeine)
2. Current serious medical illness, including migraine headaches. '
3. Currently on psychotropic medications with dosage unchanged for less than four weeks prior to study entry OR plan to make changes in medication within 2 months after starting the study
4. History of seizure except those therapeutically induced by electroconvulsive therapy (ECT), history of epilepsy in self or first degree relatives, stroke, brain surgery, head injury, cranial metal implants, known structural brain lesion, devices that may be affected by TMS (pacemaker, medication pump, cochlear implant, implanted brain stimulator).
5. Diagnosed with the following conditions: psychotic disorder, any DSM disorder secondary to a general medical condition, or substance-induced, Bipolar I disorder (current or lifetime), life-threatening anorexia or any other disorder requiring immediate hospitalization, high-risk for suicidal behavior, including current suicidal ideation with a method and plan or hospitalization for suicidal behavior within 1yr before the study.
6. Currently engaged or planning to engage in other treatment during the course of the study (including behavior therapy, or other types of individual, family, or group psychotherapy/counseling).
7. Is diagnosed with a clinically defined neurological disorder including, but not limited to: any condition likely to be associated with increased intracranial pressure; space occupying brain lesion; history of stroke, transient ischemic attack within two years; cerebral aneurysm; dementia; Parkinson's disease; Huntington's disease; Multiple sclerosis.
8. Has increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or currently taking medication that lowers the seizure threshold (e.g Wellbutrin, Adderall, Clozaril).
9. Has any of the following treatment histories: TMS treatment at any point in their lifetime; use of any investigational drug or device within 4 weeks of the screening.
10. Subjects with cochlear implants
11. Women who are pregnant or breast feeding
12. Chronic absence of shelter or impending jail that would make consistent participation in the study difficult
13. Cannot easily come to Duke several times for the study procedures
14. Does not have a mobile phone or is unwilling to use mobile phone for ambulatory assessment
15. Does not speak/understand English enough to benefit from the psychotherapeutic intervention
16. Intellectual disability

For imaging arm of the study, participants must also be able to tolerate an MRI, thus must be eligible based on the MRI safety screening form.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrada D Neacsiu, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center-Civitan Bldg, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gross, J. J. Handbook of Emotion Regulation, Second Edition. (The Guilford Press, 2013).
- [Background] Neacsiu AD, Eberle JW, Kramer R, Wiesmann T, Linehan MM. Dialectical behavior therapy skills for transdiagnostic emotion dysregulation: a pilot randomized controlled trial. Behav Res Ther. 2014 Aug;59:40-51. doi: 10.1016/j.brat.2014.05.005. Epub 2014 May 27. PMID 24974307
- [Background] Kazdin AE, Blase SL. Rebooting Psychotherapy Research and Practice to Reduce the Burden of Mental Illness. Perspect Psychol Sci. 2011 Jan;6(1):21-37. doi: 10.1177/1745691610393527. Epub 2011 Feb 3. PMID 26162113
- [Background] Luber B, Steffener J, Tucker A, Habeck C, Peterchev AV, Deng ZD, Basner RC, Stern Y, Lisanby SH. Extended remediation of sleep deprived-induced working memory deficits using fMRI-guided transcranial magnetic stimulation. Sleep. 2013 Jun 1;36(6):857-71. doi: 10.5665/sleep.2712. PMID 23729929
- [Background] Feeser M, Prehn K, Kazzer P, Mungee A, Bajbouj M. Transcranial direct current stimulation enhances cognitive control during emotion regulation. Brain Stimul. 2014 Jan-Feb;7(1):105-12. doi: 10.1016/j.brs.2013.08.006. Epub 2013 Sep 21. PMID 24095257
- [Background] Pitman RK, Orr SP, Forgue DF, de Jong JB, Claiborn JM. Psychophysiologic assessment of posttraumatic stress disorder imagery in Vietnam combat veterans. Arch Gen Psychiatry. 1987 Nov;44(11):970-5. doi: 10.1001/archpsyc.1987.01800230050009. PMID 3675137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from the community occurred between 3/1/2016 and 2/17/2019 . Additional funding was received in 2017 to collect additional data. Two conditions were added where procedures were identical but targeting for neurostimulation was done using functional neuroimaging data. Participants were recruited for both the study and the sub study and assigned to one at intake.
Pre-assignment Details: We enrolled 148 participants in both studies of which 78 were randomized in one of the two studies (main study or sub study). Twenty seven participants decided to withdraw after intake.In addition, 42 participants were excluded after enrollment (e.g., TMS was contraindicated, did not meet criteria for any DSM disorder, had current psychosis/mania/addiction, etc). One participant piloted the procedures and was also excluded from analyses.
Groups:
- Cognitive Restructuring+rTMS (Left): Participants in this arm will be administered the neuromodulation enhanced cognitive restructuring intervention over the left side of the brain and will partake in short term and long term follow up testing.
  Cognitive Restructuring: Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.The specific neurostimulation target will be established using the 10-20 system.
  rTMS: rTMS is a neurostimulation intervention where the participant receives 15 minutes of high frequency (10 HZ) transcranial magnetic stimulation pulses
- Cognitive Restructuring + Sham rTMS: Participants in this arm will receive cognitive restructuring alone as an active intervention and will partake in short term and long term follow up testing. The specific neurostimulation target will be established using the 10-20 system.
  Cognitive Restructuring: Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.
  Sham rTMS: Sham rTMS is a placebo intervention aimed to mimic the effects of repetitive transcranial magnetic stimulation with no known direct benefit for the participant.
- Cognitive Restructuring+rTMS (Right): Participants in this arm will be administered the neuromodulation enhanced cognitive restructuring intervention over the right side of the brain and will partake in short term and long term follow up testing. The specific neurostimulation target will be established using the 10-20 system.
  Cognitive Restructuring: Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.
  rTMS: rTMS is a neurostimulation intervention where the participant receives 15 minutes of high frequency (10 HZ) transcranial magnetic stimulation pulses
- Cognitive Restructuring+rTMS (Left) With Functional Targeting: Participants in this arm will be administered the neuromodulation enhanced cognitive restructuring intervention over the left side of the brain and will partake in short term and long term follow up testing. The specific neurostimulation target will be established using neuroimaging functional data.
  Cognitive Restructuring: Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.
  rTMS: rTMS is a neurostimulation intervention where the participant receives 15 minutes of high frequency (10 HZ) transcranial magnetic stimulation pulses
- Cognitive Restructuring + Sham rTMS With Functional Targeting: Participants in this arm will receive cognitive restructuring alone as an active intervention and will partake in short term and long term follow up testing.
  Cognitive Restructuring: Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.The specific neurostimulation target will be established using neuroimaging functional data.
  Sham rTMS: Sham rTMS is a placebo intervention aimed to mimic the effects of repetitive transcranial magnetic stimulation with no known direct benefit for the participant.
Period: Overall Study
Arm/Group | Cognitive Restructuring+rTMS (Left) | Cognitive Restructuring + Sham rTMS | Cognitive Restructuring+rTMS (Right) | Cognitive Restructuring+rTMS (Left) With Functional Targeting | Cognitive Restructuring + Sham rTMS With Functional Targeting
Started | 14 | 15 | 18 | 16 | 15
Completed | 11 | 14 | 15 | 14 | 11
Not Completed | 3 | 1 | 3 | 2 | 4
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Completers (i.e., those who attempted and could complete the information). Those who were intent to treat who could not tolerate the intervention are not represented in these descriptive statistics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Restructuring+rTMS (Left) | Cognitive Restructuring + Sham rTMS | Cognitive Restructuring+rTMS (Right) | Cognitive Restructuring+rTMS (Left) With Functional Targeting | Cognitive Restructuring + Sham rTMS With Functional Targeting | Total
Number analyzed (Participants) | 13 | 14 | 15 | 14 | 13 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.08 (13.77) | 29.43 (10.95) | 28.80 (7.07) | 32.64 (14.19) | 35.77 (13.50) | 31.64 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 13 | 11 | 11 | 58
  Male | 2 | 2 | 2 | 3 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 1 | 2 | 8
  Not Hispanic or Latino | 10 | 13 | 14 | 13 | 11 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 3 | 3 | 3 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 3 | 1 | 10
  White | 10 | 9 | 9 | 7 | 9 | 44
  More than one race | 0 | 0 | 1 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 14 | 15 | 14 | 13 | 69
ERQ Reappraisal Score [Mean (Standard Deviation); unit: units on a scale] — Emotion Regulation Questionnaire (ERQ). The ERQ (6) is a 10-item self-report inventory that assesses the routine use of two cognitive emotion regulation strategies: expressive suppression and cognitive reappraisal. The items use a 7-point Likert scale with responses ranging from one (strongly disagree) to 7 (strongly agree). The data reported here is for the Cognitive reappraisal subscale which can range from 1 to 7, with higher scores indicating more use of reappraisal to alter emotions.
  units on a scale | 3.26 (0.87) | 3.21 (0.76) | 3.51 (0.79) | 4.10 (1.35) | 4.44 (1.33) | 3.70 (1.12)
DERS Total Score [Mean (Standard Deviation); unit: units on a scale] — Difficulties in Emotion Regulation Scale (DERS). The DERS (49) is a 36-item self-report measure of individuals' typical levels of emotion dysregulation across six domains. Participants respond on a Likert scale ranging from 1 (almost never) to 5 (almost always). The total score ranges from 36 to 180 with higher scores indicating higher dysregulation than lower scores.
  units on a scale | 93.54 (27.55) | 118.57 (13.72) | 95.67 (19.05) | 109.57 (17.02) | 110.39 (18.54) | 105.51 (21.27)

OUTCOME MEASURES:

1. Primary Outcome: Time to Return to Heart Rate Baseline During the Regulation Period During Training
Description: The estimated marginal mean of the difference in length of time that it takes participants to reduce emotional arousal after three emotional inductions when they use Cognitive Restructuring (CR) with or without the enhancing effects of transcranial magnetic stimulation (TMS). Psychophysiological measurements were collected continuously using the BIOPAC MP-150. For each baseline, heart rate (HR) was averaged from the last 240s. Time to return to one's HR baseline was defined as the amount of time (e.g., number of seconds) it took from the beginning of regulation for the continuously monitored HR to reach a value that was lower than the average pre-stimulus baseline HR. Lower numbers indicate quicker regulation (desirable outcome). A baseline value for regulation duration was computed as the time it took during habituation for the person to return to HR baseline. Number of seconds was transformed with a logarithmic function for analyses to achieve normality.
Time Frame: 1 week after intake
Population: Each participant went through three stressor-regulation periods during the intervention. Only those who stressed at least during one of the three stressor periods were included in this analysis. Missing participants from the total ITT sample did not stress at all during the intervention stressor tasks. The results presented are estimated marginal means from the MMANOVA analysis that included this information
Measure: Least Squares Mean (Standard Error); unit: log (seconds)
Groups:
- Cognitive Restructuring+rTMS (Left): Participants in this arm will be administered the neuromodulation enhanced cognitive restructuring intervention over the left side of the brain and will partake in short term and long term follow up testing. The specific neurostimulation target will be established using the 10-20 system (i.e., scalp measurements).
  Cognitive Restructuring: Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.The specific neurostimulation target will be established using the 10-20 system.
  rTMS: rTMS is a neurostimulation intervention where the participant receives 40 minutes of high frequency (10 HZ) transcranial magnetic stimulation pulses (4 s train, 26s inter-train interval). The first 10 minutes of neurostimulation will happen during a habituation period in the absence of emotional induction and cognitive restructuring. the rest of 30 minutes will happen in chunks of 10 minutes, following a 2 minute negative emotional induction using autobiographical stressors, while the participant engages in cognitive restructuring.
- Cognitive Restructuring + Sham rTMS: Participants in this arm will receive cognitive restructuring alone as an active intervention and will partake in short term and long term follow up testing. The specific neurostimulation target will be established using the 10-20 system (i.e., scalp measurements).
  Cognitive Restructuring: Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.
  Sham rTMS: Sham rTMS is a placebo intervention aimed to mimic the effects of repetitive transcranial magnetic stimulation with no known direct benefit for the participant. Sound and scalp stimulation made the experience similar to active neurostimulation.
- Cognitive Restructuring+rTMS (Right): Participants in this arm will be administered the neuromodulation enhanced cognitive restructuring intervention over the right side of the brain and will partake in short term and long term follow up testing. The specific neurostimulation target will be established using the 10-20 system (i.e., scalp measurements).
  Cognitive Restructuring: Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.
  rTMS: rTMS is a neurostimulation intervention where the participant receives 40 minutes of high frequency (10 HZ) transcranial magnetic stimulation pulses (4 s train, 26s inter-train interval). The first 10 minutes of neurostimulation will happen during a habituation period in the absence of emotional induction and cognitive restructuring. the rest of 30 minutes will happen in chunks of 10 minutes, following a 2 minute negative emotional induction using autobiographical stressors, while the participant engages in cognitive restructuring.
- Cognitive Restructuring+rTMS (Left) With Functional Targeting: Participants in this arm will be administered the neuromodulation enhanced cognitive restructuring intervention over the left side of the brain and will partake in short term and long term follow up testing. The specific neurostimulation target will be established using neuroimaging functional data.
  Cognitive Restructuring: Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.
  rTMS: rTMS is a neurostimulation intervention where the participant receives 40 minutes of high frequency (10 HZ) transcranial magnetic stimulation pulses (4 s train, 26s inter-train interval). The first 10 minutes of neurostimulation will happen during a habituation period in the absence of emotional induction and cognitive restructuring. the rest of 30 minutes will happen in chunks of 10 minutes, following a 2 minute negative emotional induction using autobiographical stressors, while the participant engages in cognitive restructuring.
- Cognitive Restructuring + Sham rTMS With Functional Targeting: Participants in this arm will receive cognitive restructuring alone as an active intervention and will partake in short term and long term follow up testing.
  Cognitive Restructuring: Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.The specific neurostimulation target will be established using neuroimaging functional data.
  Sham rTMS: Sham rTMS is a placebo intervention aimed to mimic the effects of repetitive transcranial magnetic stimulation with no known direct benefit for the participant. A specific neurostimulation target for the sham stimulation will be established using neuroimaging functional data. Sound and scalp stimulation made the experience similar to active neurostimulation.
Arm/Group | Cognitive Restructuring+rTMS (Left) | Cognitive Restructuring + Sham rTMS | Cognitive Restructuring+rTMS (Right) | Cognitive Restructuring+rTMS (Left) With Functional Targeting | Cognitive Restructuring + Sham rTMS With Functional Targeting
Number analyzed (Participants) | 12 | 11 | 13 | 11 | 10
log (seconds) | 1.591 (.093) | 1.828 (.095) | 1.505 (.089) | 1.534475 (.154) | 1.946232 (.173)
Statistical Analysis 1: Comparison: Cognitive Restructuring + Sham rTMS vs Cognitive Restructuring+rTMS (Right); A mixed models analysis of variance (MMANOVA) examining regulation duration during each regulation period was conducted using treatment condition (active right, active left, sham), experimental condition (regulation1, regulation2, regulation3), and baseline as predictors; Test type: Superiority — Aimed to recruit 20 participants in each condition to align with other neurostimulation studies where 6-20 adults per condition were sufficient to demonstrate proof-of-concept for novel treatments (Bentwich et al., 2011; Cunningham et al., 2015); p = 0.019, Mixed Models Analysis — A priori threshold for significance was .05; Mean Difference (Net) = -0.323, 95% CI 2-sided [-.590 to -.056], Standard Error of Mean .131 — The results presented are between the active right and sham conditions
Statistical Analysis 2: Comparison: Cognitive Restructuring+rTMS (Left) vs Cognitive Restructuring + Sham rTMS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .08, Mixed Models Analysis; Mean Difference (Net) = .237, 95% CI 2-sided [-.034 to .508], Standard Error of Mean .133
Statistical Analysis 3: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; Regulation duration was transformed using a logarithmic transformation to achieve normality; Test type: Superiority; p = .033, Mixed Models Analysis — A priori threshold for significance was set to .05; we controlled for baseline and for the distance between the brain and the scalp; Mean Difference (Net) = -.227, 95% CI 2-sided [-.434 to -.020], Standard Error of Mean .103

2. Primary Outcome: Time to Return to Heart Rate Baseline During the Regulation Period at Follow up
Description: The investigators will examine difference in length of time that it takes participants to reduce emotional arousal (as measured with physiological indicators) after an emotional induction when they use CR. This measure, was collected at the 1 month follow up assessment. Only one stressor-regulation period was presented at follow up. The number of seconds it took for participants to return to the pre-stimulus baseline during the regulation period was transformed with a log function for normality. Lower numbers indicate quicker regulation, a desirable outcome.
Time Frame: 1 month
Population: only participants who "stressed" during the follow up stressor task (i.e., their heart rate was above baseline at the beginning of the follow up regulation period) were included in these analyses. Missing participants did not stress at follow up.
Measure: Mean (Standard Error); unit: log (seconds)
Arm/Group | Cognitive Restructuring+rTMS (Left) | Cognitive Restructuring + Sham rTMS | Cognitive Restructuring+rTMS (Right) | Cognitive Restructuring+rTMS (Left) With Functional Targeting | Cognitive Restructuring + Sham rTMS With Functional Targeting
Number analyzed (Participants) | 8 | 9 | 10 | 9 | 5
log (seconds) | 1.448 (0.089) | 1.286 (0.062) | 1.1474 (0.110) | 1.5535 (0.0936) | 1.4055 (0.14923)
Statistical Analysis 1: Comparison: Cognitive Restructuring+rTMS (Left) vs Cognitive Restructuring + Sham rTMS; A univariate general linear model was employed to test of regulation duration, transformed for normality; Test type: Superiority; p = .51, ANOVA — A priori set threshold for statistical significance was 0.05; Mean Difference (Net) = -.124, 95% CI 2-sided [-0.504 to .256], Standard Error of Mean 0.184
Statistical Analysis 2: Comparison: Cognitive Restructuring + Sham rTMS vs Cognitive Restructuring+rTMS (Right); Test type: Superiority; p = .97, ANOVA; Mean Difference (Net) = .007, 95% CI 2-sided [-.364 to .378], Standard Error of Mean .180
Statistical Analysis 3: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; A t test of the variable 'time it took to return to HR baseline', transformed for normality was used to examine between condition differences at the 1 month follow up; Test type: Superiority; p = 0.39, t-test, 2 sided — A priori set significance threshold was 0.05; Mean Difference (Net) = 0.147993, 95% CI 2-sided [-0.215936 to 0.511921], Standard Error of Mean 0.167031

3. Primary Outcome: Physiological Emotion Regulation
Description: The investigators will record heart rate continuously throughout the intervention and then extract high frequency heart rate variability (an index of emotion regulation) from the regulation periods. Continuously recorded HR was divided into 120 s bins, and HF-HRV was extracted from cleaned raw ECG from each bin. Baseline HF-HRV was measured at the beginning of the experiment and right before each autobiographical stressor presentation. The treatment condition (active left, active right, or sham), baselines, the experimental condition (regulation 1, 2, and 3), and the time within each experimental condition (0 to 4 for each 120 s segment within that period) were used to predict HF-HRV. Higher HF-HRV indicates enhanced regulation, a desirable outcome. To make interpretation easier, the raw HF-HRV score was multiplied with 1000000. To achieve normality, this multiplied score was transformed with a logarithmic function.
Time Frame: 1 week after study start
Measure: Least Squares Mean (Standard Error); unit: lg(1000000*milliseconds)
Groups:
- Cognitive Restructuring+rTMS (Left): Participants in this arm will be administered the neuromodulation enhanced cognitive restructuring intervention over the left side of the brain and will partake in short term and long term follow up testing.
  Cognitive Restructuring: Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.The specific neurostimulation target will be established using the 10-20 system.
  rTMS: rTMS is a neurostimulation intervention where the participant receives 10 minutes of high frequency (10 HZ) transcranial magnetic stimulation pulses (4s train 26 s inter train interval). the 10-minute administration was repeated 4 times
- Cognitive Restructuring+rTMS (Right): Participants in this arm will be administered the neuromodulation enhanced cognitive restructuring intervention over the right side of the brain and will partake in short term and long term follow up testing. The specific neurostimulation target will be established using the 10-20 system.
  Cognitive Restructuring: Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.
  rTMS: rTMS is a neurostimulation intervention where the participant receives 10 minutes of high frequency (10 HZ) transcranial magnetic stimulation pulses. (4s train 26 s inter train interval). the 10-minute administration was repeated 4 times
- Cognitive Restructuring+rTMS (Left) With Functional Targeting: Participants in this arm will be administered the neuromodulation enhanced cognitive restructuring intervention over the left side of the brain and will partake in short term and long term follow up testing. The specific neurostimulation target will be established using neuroimaging functional data.
  Cognitive Restructuring: Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal. Specifically, participants learn how to distance themselves from the situation, think of the memory as just a memory, or focus on alternative explanations or facets of the situation that are less emotionally upsetting.
  rTMS: rTMS is a neurostimulation intervention where the participant receives 10 minutes of high frequency (10 HZ) transcranial magnetic stimulation pulses. (4s train 26 s inter train interval). the 10-minute administration was repeated 4 times
Arm/Group | Cognitive Restructuring+rTMS (Left) | Cognitive Restructuring + Sham rTMS | Cognitive Restructuring+rTMS (Right) | Cognitive Restructuring+rTMS (Left) With Functional Targeting | Cognitive Restructuring + Sham rTMS With Functional Targeting
Number analyzed (Participants) | 13 | 14 | 15 | 14 | 13
lg(1000000*milliseconds) | 1.919 (.041) | 1.763 (.039) | 1.869 (.038) | 1.722 (.016) | 1.549 (.017)
Statistical Analysis 1: Comparison: Cognitive Restructuring+rTMS (Left) vs Cognitive Restructuring + Sham rTMS; In the original study (CR+active left rTMS vs CR+ active right rTMS vs CR+sham rTMS), mixed-effects hierarchical linear models (MMANOVA) with analytically determined covariance structures were used to analyze the repeated measures data. We hypothesized that active neurostimulation would increase HF-HRV during regulation; Test type: Superiority — HF-HRV was transformed using the function lg10*(HF-HRV*1000000) in order to be normally distributed; p = .022, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = .16, 95% CI 2-sided [.044 to .267], Standard Deviation .51
Statistical Analysis 2: Comparison: Cognitive Restructuring + Sham rTMS vs Cognitive Restructuring+rTMS (Right); MMANOVA; Test type: Superiority; p = 0.0499, Mixed Models Analysis; Mean Difference (Net) = .11, 95% CI 2-sided [0.000037 to 0.213074], Standard Error of Mean .052
Statistical Analysis 3: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; In the supplemental study (CR+active left rTMS with functional targeting vs CR+sham rTMS), mixed-effects hierarchical linear models (MMANOVA) with analytically determined covariance structures were used to analyze the repeated measures data. We hypothesized that active neurostimulation would increase HF-HRV during regulation when compared with sham; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < .000001, Mixed Models Analysis — Significance threshold was set at p = 0.05; Mean Difference (Net) = .172, 95% CI 2-sided [.129 to .215], Standard Deviation .38 — The MMANOVA analysis used an unstructured covariance structure

4. Primary Outcome: Changes in Activation in the Neural Emotion Regulation Network
Description: For groups 4 &5, the investigators collected functional imaging data while participants engaged in an emotion regulation task. We examined the BOLD response change in the contrast between down-regulating negative emotions and feeling negative emotions a week after intervention controlling for the maximum change in this contrast at intake. Specifically we examined changes in activation in the dorsolateral prefrontal cortex (dlPFC), ventrolateral PFC (vlPFC), ventromedial PFC (vmPFC), the amygdala and insula. Data were first preprocessed with fMRIprep and MRIQC. At the first level, functional data were analyzed as individual runs, using a general linear model (GLM) in which trial events were convolved with a double-gamma hemodynamic response function. The [Restructure- Feel_negative] contrast was then used to generate Level 2 analysis, in which BOLD activity for each of the four runs were combined using a fixed-effect model. Higher numbers indicate more activation (desired outcome).
Time Frame: 1 week
Population: This data was not collected from all participants. It was only collected for a subset of participants assigned to the imaging sub study (groups 4 and 5). The numbers presented represent estimated marginal means from the MANCOVA analysis comparing conditions and covarying maximum activation within the contrast at intake.
Measure: Least Squares Mean (Standard Error); unit: Maximum % signal change in ROI
Arm/Group | Cognitive Restructuring+rTMS (Left) | Cognitive Restructuring + Sham rTMS | Cognitive Restructuring+rTMS (Right) | Cognitive Restructuring+rTMS (Left) With Functional Targeting | Cognitive Restructuring + Sham rTMS With Functional Targeting
Number analyzed (Participants) | 0 | 0 | 0 | 13 | 13
Maximum % signal change in ROI
  dlPFC |  |  |  | 0.573 (.065) | .462 (.065)
  vlPFC |  |  |  | 0.965 (0.102) | 0.606 (0.102)
  vmPFC |  |  |  | 2.597 (0.326) | 2.376 (0.326)
  amygdala |  |  |  | 0.664 (0.125) | 0.485 (0.125)
  Insula |  |  |  | .543 (0.05) | .522 (0.05)
Statistical Analysis 1: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; Difference between treatment conditions in dlPFC activation change between feeling negative emotions and downregulation of negative affect a week after intervention, when controlling for baseline activation difference; Test type: Superiority; p = .236, ANCOVA — A priori threshold was set to 0.05; Brain to skull difference and intake difference in dlPFC activation between regulation and feeling negative were included as confounds; Mean Difference (Net) = .111, 95% CI 2-sided [-0.078086 to 0.300661], Standard Error of Mean 0.091544 — Parameter estimate is the value of the difference between active stimulation and sham stimulation
Statistical Analysis 2: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; Expected significantly higher activation following active intervention in the vlPFC when compared to sham when engaging in downregulation versus passive experience of negative emotions induced with autobiographical stressors. ROI data was extracted using FSL featquery. A univariate general linear model excluding one outlier from the active condition was conducted for this outcome measure; Test type: Superiority; p = 0.020347, ANCOVA — Threshold was set at 0.05 a priori; Brain to skull difference and intake difference in vlpfc activation between regulation and feeling negative were included as confounds; Mean Difference (Net) = 0.359024, 95% CI 2-sided [0.061000 to 0.657049], Standard Error of Mean 0.144067
Statistical Analysis 3: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; Expected significantly higher activation following active intervention in the vmPFC when compared to sham when engaging in downregulation versus passive experience of negative emotions induced with autobiographical stressors. ROI data was extracted with FSL featquery; Test type: Superiority; p = 0.635, ANCOVA — A priori threshold was set to .05; Brain to skull difference and intake difference in vmpfc activation between regulation and feeling negative were included as confounds; Mean Difference (Net) = 0.221683, 95% CI 2-sided [-0.732963 to 1.176330], Standard Error of Mean 0.461481
Statistical Analysis 4: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; Expected significantly lower activation following active intervention in the amygdala when compared to sham when engaging in downregulation versus passive experience of negative emotions induced with autobiographical stressors. ROI data was extracted with featquery (FSL); Test type: Superiority; p = .324, ANCOVA — a priori set threshold was 0.05; Brain to skull difference and intake difference in amygdala activation between regulation and feeling negative were included as confounds; Mean Difference (Net) = 0.179412, 95% CI 2-sided [-0.188868 to 0.547692], Standard Error of Mean 0.178029
Statistical Analysis 5: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; Expected significantly lower activation following active intervention in the insula when compared to sham when engaging in downregulation versus passive experience of negative emotions induced with autobiographical stressors. FSL featquery tool was used to extract ROI (region of interest) data; Test type: Superiority; p = 0.768190, ANCOVA — A priori set threshold was 0.05; Brain to skull difference and intake difference in insula activation between regulation and feeling negative were included as confounds; Mean Difference (Net) = 0.021231, 95% CI 2-sided [-0.126027 to 0.168489], Standard Error of Mean 0.071185

5. Secondary Outcome: Acceptability, as Measured by Qualitative Exit Interview
Description: The investigators will examine how acceptable participants find the intervention. A previously developed in-house interview (A. D. Neacsiu, Luber, et al., 2018) was administered at the 1-month follow up, and it included Likert-type questions about feasibility, acceptability, and overall satisfaction rated on a scale from 0 (not at all) to 9 (extremely; secondary outcomes).
Time Frame: 1 month
Population: Only participants who were not lost to contact by the last session of the study provided data for this outcome measure. One participant did not complete the acceptability portion of the exit interview and as a result their data cannot be included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Restructuring+rTMS (Left) | Cognitive Restructuring + Sham rTMS | Cognitive Restructuring+rTMS (Right) | Cognitive Restructuring+rTMS (Left) With Functional Targeting | Cognitive Restructuring + Sham rTMS With Functional Targeting
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 11
units on a scale | 7.11 (1.07) | 7.48 (0.92) | 7.20 (1.34) | 6.99 (1.25) | 7.65 (0.91)
Statistical Analysis 1: Comparison: Cognitive Restructuring+rTMS (Left) vs Cognitive Restructuring + Sham rTMS; Likert-type questions about acceptability were rated on a scale from 0 (not at all) to 9 (extremely) and then averaged to create a mean for acceptability. This average score was normally distributed and therefore was entered into a univariate general linear model where acceptability was entered as a dependent variable and condition as a fixed factor; Test type: Superiority; p = 0.69, ANOVA — a priori threshold for significance was 0.05; Mean Difference (Net) = .37, 95% CI 2-sided [-0.553 to 1.293], Standard Error of Mean .455
Statistical Analysis 2: Comparison: Cognitive Restructuring + Sham rTMS vs Cognitive Restructuring+rTMS (Right); Test type: Superiority; p = .53, ANOVA; Mean Difference (Net) = .27, 95% CI 2-sided [-.592 to 1.139], Standard Error of Mean .43
Statistical Analysis 3: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; we compared differences in acceptability between conditions using an independent samples t-test (acceptability was normally distributed); Test type: Superiority; p = 0.15, t-test, 2 sided — a priory threshold for significance was .05; Mean Difference (Net) = -.66, 95% CI 2-sided [-1.59 to 0.27], Standard Error of Mean .45

6. Secondary Outcome: Feasibility, as Measured by Qualitative Exit Interview
Description: The investigators will examine how feasible the proposed intervention is. A previously developed in-house interview (A. D. Neacsiu, Luber, et al., 2018) was administered at the 1-month follow up, and it included Likert-type questions about feasibility, acceptability, and overall satisfaction rated on a scale from 0 (not at all) to 9 (extremely; secondary outcomes).
Time Frame: 1 month
Population: Only participants who were not lost to contact by the last study session provided data for this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Restructuring+rTMS (Left) | Cognitive Restructuring + Sham rTMS | Cognitive Restructuring+rTMS (Right) | Cognitive Restructuring+rTMS (Left) With Functional Targeting | Cognitive Restructuring + Sham rTMS With Functional Targeting
Number analyzed (Participants) | 11 | 14 | 15 | 14 | 11
units on a scale | 6.4545 (0.83) | 6.7500 (0.87) | 6.7481 (0.555) | 6.3651 (0.886) | 6.4646 (0.9645)
Statistical Analysis 1: Comparison: Cognitive Restructuring+rTMS (Left) vs Cognitive Restructuring + Sham rTMS; We compared differences between conditions in the perceived feasibility of the procedures. Feasibility average was normally distributed and therefore a general linear model, univariate was employed to test between condition effects; Test type: Superiority; p = 0.551, ANOVA — a priori threshold was set to 0.05; Mean Difference (Net) = 0.295, 95% CI 2-sided [-0.322 to 0.912], Standard Error of Mean 0.304
Statistical Analysis 2: Comparison: Cognitive Restructuring + Sham rTMS vs Cognitive Restructuring+rTMS (Right); Test type: Superiority; p = .995, ANOVA; Mean Difference (Net) = 0.002, 95% CI 2-sided [-.567 to .571], Standard Error of Mean 0.281
Statistical Analysis 3: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; We examined differences in feasibility between the active and sham condition in the sub-study where fMRI targeting was utilized. Average feasibility was normally distributed and therefore an independent samples t-test was used to test this outcome; Test type: Superiority; p = 0.791, t-test, 2 sided — A priori threshold for statistical significance was set to 0.05; df = 23; Mean Difference (Net) = -0.09957, 95% CI 2-sided [-0.8672 to 0.6681], Standard Error of Mean 0.371

7. Secondary Outcome: Change in General Psychological Distress, as Measured by the Outcome Questionaire -45
Description: The investigators will examine change in general psychological distress after the intervention. The Outcome Questionnaire-45 (OQ-45) is a 45-item self-report measure used to track severity of psychopathology throughout treatment. It consists of subscales that identify three types of problems that lead to general stress: psychological symptoms, interpersonal conflicts, and problems with social roles. Items are rated on a Likert scale ranging from 0 (never) to 4 (almost always). We computed the total score (ranging from 0 to 180) from data collected at intake, at 1 week after the intervention, and at 1 month after the intervention. Higher score indicate higher psychopathological distress than lower scores. The estimated marginal means from the growth model comparing differences between conditions are presented in the table below.
Time Frame: 1 week and 1 month
Population: Only participants who provided data were included. In the first study (first 3 groups) one participant from the active right condition did not complete the 1-week follow-up self-reports. One sham, three active left, and one active right participant could not tolerate the intervention and dropped. In the second study (last 2 groups) two participants could not tolerate the intervention and dropped in each condition. One participant in sham did not complete his OQ-45 measure at follow up.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Restructuring+rTMS (Left) | Cognitive Restructuring + Sham rTMS | Cognitive Restructuring+rTMS (Right) | Cognitive Restructuring+rTMS (Left) With Functional Targeting | Cognitive Restructuring + Sham rTMS With Functional Targeting
Number analyzed (Participants) | 13 | 14 | 14 | 14 | 12
score on a scale | 59.996 (5.48) | 53.955 (5.29) | 53.049 (5.06) | 74.41 (5.45) | 63.95 (5.73)
Statistical Analysis 1: Comparison: Cognitive Restructuring+rTMS (Left) vs Cognitive Restructuring + Sham rTMS; To test the long-term effects of the intervention, a MMANOVA model was conducted examining between-condition differences at the 1-week and 1-month follow-up in the OQ-45. Baseline was co-varied; Test type: Superiority; p = 0.61, Mixed Models Analysis — A priori threshold was set to 0.05; Mean Difference (Net) = 6.04, 95% CI 2-sided [-9.522964 to 21.604620], Standard Error of Mean 8.048
Statistical Analysis 2: Comparison: Cognitive Restructuring + Sham rTMS vs Cognitive Restructuring+rTMS (Right); Test type: Superiority; p = .90, Mixed Models Analysis — a priori threshold was set to .05; Mean Difference (Net) = -.906, 95% CI 2-sided [-15.83 to 14.02], Standard Error of Mean 7.37
Statistical Analysis 3: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; Test type: Superiority; p = .20, Mixed Models Analysis — threshold was set to 0.05 a priori; Mean Difference (Net) = 10.46, 95% CI 2-sided [-5.971581 to 26.892619], Standard Error of Mean 7.93 — HLM models used a compound symmetry covariance structure

8. Secondary Outcome: Change in Daily General Emotional Distress
Description: The investigators will examine change in emotional distress after the intervention as measured by daily mobile phone ratings 8 times/day for 7 days of subjective units of distress; SUDS). The 8 ratings/day will then be averaged into a mean/day. This daily SUDS mean (range 0-9) will be entered in analyses. Higher SUDS indicates more distress.
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: units on a scale per day
Arm/Group | Cognitive Restructuring+rTMS (Left) | Cognitive Restructuring + Sham rTMS | Cognitive Restructuring+rTMS (Right) | Cognitive Restructuring+rTMS (Left) With Functional Targeting | Cognitive Restructuring + Sham rTMS With Functional Targeting
Number analyzed (Participants) | 13 | 14 | 15 | 14 | 13
units on a scale per day | 1.388 (0.217) | 1.941 (0.212) | 1.791 (0.205) | 2.026 (0.269) | 1.395 (0.293)
Statistical Analysis 1: Comparison: Cognitive Restructuring+rTMS (Left) vs Cognitive Restructuring + Sham rTMS vs Cognitive Restructuring+rTMS (Right); Hypothesized that active neurostimulation would lead to lower daily distress than sham stimulation. We used a hierarchical linear model (HLM) for this analysis with an identity covariance structure (random intercept and random slope); Test type: Superiority; p = .034, Mixed Models Analysis — A priori threshold was set to .05 for significance; Subjective Units of Distress (SUDS) right before the intervention were co-varied as baseline; Mean Difference (Net) = -0.55, 95% CI 2-sided [-1.062356 to -0.043203], Standard Error of Mean 0.258 — Results reported are for active left vs. sham comparison
Statistical Analysis 2: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; Hypothesized that active neurostimulation will lead to less daily distress than sham neurostimulation during the ambulatory data collection. An HLM analysis was conducted using an unstructured covariance structure and reported distress right before the intervention as baseline; Test type: Superiority; p = .133, Mixed Models Analysis — A priori set threshold was .05; Mean Difference (Net) = 0.631, 95% CI 2-sided [-.208 to 1.47], Standard Error of Mean 0.404

9. Secondary Outcome: Change in Emotion Dysregulation and Functional Impairment
Description: The investigators will examine changes in the reappraisal scale of the Emotion Regulation Questionnaire (ERQ; range 1-7), in the total score from the Difficulties with Emotion Regulation Scale (DERS; range 36-180), and in the total score from the work and social adjustment functional impairment scale (WSAS; range 0-40) from before to after the one time intervention. Higher ERQ-Reappraisal scores indicate more use of cognitive restructuring (a favorable outcome). Lower DERS total score and lower WSAS average score indicate lower overall emotional dysregulation and lower impairment in functioning, which are desirable outcomes. Outcomes were analyzed using HLM models and the data presented below represents the estimate marginal means for each condition for the growth in each outcome controlling for baseline.
Time Frame: 1 week and 1 month after the intervention
Population: Only participants who provided data were included. In the first study (first 3 groups) one participant from the active right condition did not complete the 1-week follow-up self-reports. One sham, three active left, and one active right participant could not tolerate the intervention and dropped. In the second study (last 2 groups) two participants could not tolerate the intervention and dropped in each condition. One participant in sham did not complete his self-report measures at follow up.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Restructuring+rTMS (Left) | Cognitive Restructuring + Sham rTMS | Cognitive Restructuring+rTMS (Right) | Cognitive Restructuring+rTMS (Left) With Functional Targeting | Cognitive Restructuring + Sham rTMS With Functional Targeting
Number analyzed (Participants) | 13 | 14 | 14 | 14 | 12
score on a scale
  Difficulties in emotion regulation total score | 88.413631 (6.419510) | 89.341540 (6.497500) | 79.212163 (5.890947) | 99.447060 (86.259744) | 4.289242 (4.489399)
  ERQ-Reappraisal | 4.493290 (0.20) | 4.777880 (0.19) | 4.795426 (0.19) | 4.838261 (0.267571) | 4.741542 (0.281177)
  Work and Social Functioning Impairment | 12.176969 (1.941534) | 10.876197 (1.834403) | 11.853591 (1.849822) | 14.255798 (2.290357) | 10.963661 (2.295986)
Statistical Analysis 1: Comparison: Cognitive Restructuring+rTMS (Left) vs Cognitive Restructuring + Sham rTMS; Mixed model analyses of variance (MMANOVAs) were conducted to explore the difference between active and sham neurostimulation on self reported indices of regulation and psychopathology. We expected active neurostimulation to lead to less functional impairment than sham neurostimulation; Test type: Superiority; p = 0.629061, Mixed Models Analysis — A priori threshold was set to .05; Intake values for the dependent measures were covaried. The time by condition interaction term was included; Mean Difference (Net) = -1.300772, 95% CI 2-sided [-6.708548 to 4.107], Standard Error of Mean 2.670936
Statistical Analysis 2: Comparison: Cognitive Restructuring + Sham rTMS vs Cognitive Restructuring+rTMS (Right); We expected lower functional impairment in the active right versus the sham condition; Test type: Superiority; p = 0.71, Mixed Models Analysis; Mean Difference (Net) = -0.977394, 95% CI 2-sided [-6.255223 to 4.300434], Standard Error of Mean 2.605189
Statistical Analysis 3: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; Mixed model analyses of variance (MMANOVAs) were conducted to explore the difference between active and sham neurostimulation on self reported indices of regulation and psychopathology in the substudy also. We expected active neurostimulation to lead to less impairment than sham neurostimulation; Test type: Superiority; p = 0.331, Mixed Models Analysis — A priori set threshold was .05; Baseline WSAS was covaried; Mean Difference (Net) = -3.292137, 95% CI 2-sided [-10.157811 to 3.573537], Standard Error of Mean 3.314194 — The analysis compared sham versus active stimulation
Statistical Analysis 4: Comparison: Cognitive Restructuring+rTMS (Left) vs Cognitive Restructuring + Sham rTMS; Mixed model analyses of variance (MMANOVAs) were conducted to explore the difference between active and sham neurostimulation on self reported indices of regulation and psychopathology. We expected active neurostimulation to lead to more use of cognitive restructuring than sham neurostimulation; Test type: Superiority; p = 0.31, Mixed Models Analysis — A priori set threshold for significance was 0.05; baseline was covaried; Mean Difference (Net) = 0.284589, 95% CI 2-sided [-0.276030 to 0.845209], Standard Error of Mean 0.276698
Statistical Analysis 5: Comparison: Cognitive Restructuring + Sham rTMS vs Cognitive Restructuring+rTMS (Right); We hypothesized that active right neurostimulation would yield lower emotional dysregulation after the intervention when compared to sham neurostimulation; Test type: Superiority; p = 0.275257, Mixed Models Analysis; Mean Difference (Net) = 10.129377, 95% CI 2-sided [-8.394724 to 28.653479], Standard Error of Mean 9.150339
Statistical Analysis 6: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; Mixed model analyses of variance (MMANOVAs) were conducted to explore the difference between active and sham neurostimulation on self reported indices of regulation and psychopathology. We expected active neurostimulation to lead to less emotional dysregulation than sham neurostimulation; Test type: Superiority; p = 0.044, Mixed Models Analysis — A priori set significance threshold was 0.05; Mean Difference (Net) = -13.187, 95% CI 2-sided [-26.002351 to -0.372281], Standard Error of Mean 6.212753
Statistical Analysis 7: Comparison: Cognitive Restructuring+rTMS (Left) vs Cognitive Restructuring + Sham rTMS; We expected active stimulation to lead to less emotional dysregulation than sham neurostimulation. A MMANOVA model was employed, controlling for baseline; Test type: Superiority; p = .924, Mixed Models Analysis — A priori set threshold for statistical significance was 0.05; baseline was covaried; Mean Difference (Net) = 0.927909, 95% CI 2-sided [-18.508252 to 20.364071], Standard Error of Mean 9.603423
Statistical Analysis 8: Comparison: Cognitive Restructuring + Sham rTMS vs Cognitive Restructuring+rTMS (Right); we expected more use of cr following active right neurostimulation then after following sham neurostimulation; Test type: Superiority; p = .95, Mixed Models Analysis; Mean Difference (Net) = -0.017547, 95% CI 2-sided [-0.560994 to 0.525901], Standard Error of Mean 0.267983
Statistical Analysis 9: Comparison: Cognitive Restructuring+rTMS (Left) With Functional Targeting vs Cognitive Restructuring + Sham rTMS With Functional Targeting; [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p = .806, Mixed Models Analysis — A priori set significance threshold was 0.05; Baseline use of cognitive restructuring was covaried; Mean Difference (Net) = -0.096719, 95% CI 2-sided [-0.900919 to 0.707481], Standard Error of Mean 0.389897

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant throughout their participation in the study (approximately 1-2 months/participant). Adverse event data was collected starting after signing consent through completion of the follow-up final visit- about a 1-2 month time frame for each individual. If an individual was lost to contact or dropped, AE data collection ended at that point. Once the individual completed the study, AE data was no longer collected.
Arm/Group | Cognitive Restructuring+rTMS (Left) | Cognitive Restructuring + Sham rTMS | Cognitive Restructuring+rTMS (Right) | Cognitive Restructuring+rTMS (Left) With Functional Targeting | Cognitive Restructuring + Sham rTMS With Functional Targeting
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/18 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/18 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 9/14 | 6/15 | 10/18 | 9/16 | 5/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Restructuring+rTMS (Left) (N=14) | Cognitive Restructuring + Sham rTMS (N=15) | Cognitive Restructuring+rTMS (Right) (N=18) | Cognitive Restructuring+rTMS (Left) With Functional Targeting (N=16) | Cognitive Restructuring + Sham rTMS With Functional Targeting (N=15)
Manic like mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — right after neurostimulation felt good and slept about 8 hours that night. The next day began feeling more euphoric and had difficulty sleeping for the next 5 nights. She reported increased goal directed activity, and racing thoughts.
Scalp Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 6 (6) | 8 (8) | 7 (7) | 3 (3)
Increased Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncopal episode (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
mild hearing impairment (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — before intervention reported no hearing impairment but post reported mild temporary hearing impairment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT02573246/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT02573246/ICF_001.pdf